CLINICAL TRIAL: NCT07405086
Title: Knight Cancer Institute Study of Histology-Agnostic Immunotherapy With Focus on Timing: - Knight SHIFT - A Prospective, Multi-Histology Pragmatic Study
Brief Title: Morning Versus Afternoon Administration of Immunotherapy for the Treatment of Advanced or Metastatic Solid Tumors, The Knight SHIFT Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rajat Thawani, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00029305; NCI-2026-00433 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00029305 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Biliary Tract Carcinoma; Advanced Head and Neck Squamous Cell Carcinoma; Advanced Hepatocellular Carcinoma; Advanced Lung Non-Small Cell Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Melanoma; Advanced Renal Cell Carcinoma; Metastatic Biliary Tract Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hepatocellular Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Renal Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Lung Neoplasms | interventions — Specimen Handling; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (AM cohort) (Experimental): Patients receive standard of care immunotherapy before 10:30 for 4 doses in the absence of disease progression or unacceptable toxicity. Subsequent doses may be given per standard of care timing. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Immune Checkpoint Inhibitor
- Treatment (PM cohort) (Experimental): Patients receive standard of care immunotherapy after 13:30 for 4 doses in the absence of disease progression or unacceptable toxicity. Subsequent doses may be given per standard of care timing. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Immune Checkpoint Inhibitor

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Immune Checkpoint Inhibitor — Receive immune checkpoint inhibitor therapy
  Other Names: ICI

SUMMARY:
This phase IV trial is evaluating whether morning versus afternoon administration of standard of care immunotherapy impacts its effectiveness in treating patients with solid tumors that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). Immunotherapy with monoclonal antibodies may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. Circadian rhythm refers to the internal biological clock in which various processes in the body, including immune cell activity, are controlled by the time of day. Exactly how this works is not fully understood, and the researchers want to see if circadian rhythm control of the immune system can influence response to immunotherapy based on whether it is given in the morning (before 11:00 am) or afternoon (12:00pm). The time of day that immunotherapy is given (morning versus afternoon) may impact the effectiveness in treating patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival among participants receiving immunotherapy based on time of day (ToD) administration (early versus [vs.] late).

SECONDARY OBJECTIVES:

I. To compare overall survival among participants receiving immunotherapy based on ToD administration (am vs. pm).

II. To compare rates of significant immune-related adverse events (irAEs) based on ToD administration (am vs. pm).

EXPLORATORY OBJECTIVES:

I. To compare objective responses among participants receiving immunotherapy based on ToD administration (am vs. pm).

II. To compare disease control among participants receiving immunotherapy based on ToD administration (am vs. pm).

III. To compare the duration of response among participants receiving immunotherapy based on ToD administration (am vs. pm).

OUTLINE: Patients are randomized to 1 of 2 cohorts.

AM COHORT: Patients receive standard of care immunotherapy before 10:30 for 4 doses in the absence of disease progression or unacceptable toxicity. Subsequent doses may be given per standard of care timing. Patients also undergo blood sample collection throughout the study.

PM COHORT: Patients receive standard of care immunotherapy after 13:30 for 4 doses in the absence of disease progression or unacceptable toxicity. Subsequent doses may be given per standard of care timing. Patients also undergo blood sample collection throughout the study.

After completion of immunotherapy treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent before any study-specific procedures or interventions are performed
* Aged ≥ 18 years
* Histologically confirmed advanced/metastatic solid tumor as follows:

  * Non small cell lung cancer (NSCLC) (driver-negative, immune checkpoint inhibitor [ICI]-eligible)
  * Recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) (platinum-eligible),
  * Renal cell carcinoma (RCC)
  * Biliary-tract cancer (BTC)
  * Hepatocellular carcinoma (HCC)
  * Melanoma
* Planned to receive a Food and Drug Administration (FDA)-approved immune check point inhibitor (e.g., anti-PD-1, anti-PD-L1, anti-CTLA4) regimen for the treatment of their malignancy
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

Exclusion Criteria:

* Prior ICI-based regimen for treatment of cancer
* Current or prior use of immunosuppressive medication within 28 days before planned standard-of-care immunotherapy infusion, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses not exceeding 10 mg/day of prednisone (or equivalent corticosteroid)
* Uncontrolled autoimmune disease requiring immunosuppression
* Active, uncontrolled central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization to date of first progression or death (any cause), whichever occurs first (up to 2 years from date of last dose of standard-of-care immune checkpoint inhibitor [ICI])
  The associated 95% confidence interval (CI) for each treatment group will be estimated using the Kaplan-Meier method. The stratified hazard ratio (HR) and its 95% CI will be estimated using a Cox proportional-hazard model with treatment group as the independent variable and stratified by the same randomization stratification factors as were used for the log-rank test.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death (any cause) up to 2 years from date of last dose of standard-of-care ICI
  The median duration of OS and the associated 95% CI for each treatment group will be estimated using the Kaplan-Meier method. The stratified HR and its 95% CI will be estimated using a Cox proportional-hazard model with treatment group as the independent variable and stratified by the same randomization stratification factors as were used for the log-rank test.
Incidence of immune related adverse event (irAE) related time to treatment discontinuation | From date of first dose of standard-of-care ICI to date of last dose of standard-of-care ICI (an average of 2 years).
  Will be analyzed for all evaluable patients using a Kaplan-Meyer survival analysis. The number of events, percentiles for the time to discontinuation for irAE-related reasons (25%, 50% (median), and 75% percentiles), and the proportion of participants who discontinued standard-of-care for irAE-related reasons will be summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Thawani, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States